CLINICAL TRIAL: NCT04171258
Title: A Multi-center, Double-blind, Randomized, Parallel, Active-controlled, Phase I Clinical Trial to Compare the Safety and Efficacy of Botulax® Versus Botox® in Patients With Cervical Dystonia
Brief Title: Clinical Trial to Compare the Safety and Efficacy of Botulax® Versus Botox® in Patients With Cervical Dystonia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hugel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HG-BOTCD-PI-01
Record Dates: First submitted 2019-06-20; First posted 2019-11-20 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2021-11

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulax® (Experimental)
  Interventions: Drug: Botulinum toxin type A injection
- Botox® (Active Comparator)
  Interventions: Drug: Botulinum Toxin Type A Injection [Botox]

INTERVENTIONS:
Drug: Botulinum toxin type A injection — Experimental
  Other Names: Botulax®
  Arms: Botulax®
Drug: Botulinum Toxin Type A Injection [Botox] — Active Comparator
  Other Names: Botox®
  Arms: Botox®

SUMMARY:
To determine the efficacy and safety of Botulax® in treatment of cervical dystonia

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of aged over 19 years
2. Subjects diagnosed with primary cervical dystonia

Exclusion Criteria:

1. Subjects who have administered botulinum toxin within 16 weeks at the time of baseline
2. Pregnant or nursing
3. Females or males who do not agree on proper contraceptive measure

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
rate of adverse event | 12 weeks (during the clinical trial)
  To assess severity and frequency of reported adverse events and clinically-relevant changes in laboratory testing after investigational product injection.
Change From Baseline in the Total Score of the TWSTRS score. | Baseline to Week 4 , Week 8, Week 12
  The average of the change from baseline in TWSTRS-total score at Weeks 4, 8 and 12 will be determined.
  full name of TWSTRS is Toronto Western Spasmodic Torticollis Rating Scale. The validated assessment scale TWSTRS is consists of 3 sub-scales.
  1. severity (0~35 points)
  2. pain (0~20 points)
  3. disability( 0~30 points) Total score ranges from 0 to 85 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Hugel, Seoul, South Korea